CLINICAL TRIAL: NCT07247071
Title: Modifiable Risk Factors for Non-traumatic Subconjunctival Hemorrhage
Acronym: Modifiable Ris
Status: Completed | Type: Observational
Sponsor: Hallym University Kangnam Sacred Heart Hospital (Other)
Responsible Party: Principal Investigator, Young Joo Shin, Professor, Hallym University Kangnam Sacred Heart Hospital
Other Study IDs: 2023-12-01
Record Dates: First submitted 2025-11-19; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-10

CONDITIONS: Subconjunctival Hemorrhage
Keywords: Subconjunctival Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 67 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient assessments included the same systemic variables: sex, diabetes mellitus, hypertension, anti: Patient assessments included the same systemic variables: sex, diabetes mellitus, hypertension, anticoagulant use (including both antiplatelet agents and novel oral anticoagulants [NOACs]), circulatory agents, and omega-3 supplementation. Circulatory agents included Ginkgo biloba extract formulations such as Gingkomin Tab and Ginexin-F, as well as magnesium, calcium supplements, and vasodilators such as trimetazidine and limaprost.12, 13 Patients were also asked to complete structured questionnaires addressing eye rubbing, sleep deprivation, fatigue, and increased intra-abdominal pressure due to physical factors such as heavy lifting, constipation, coughing, and prone positioning. Ophthalmologic examinations were performed using fundus photography to detect retinal hemorrhages and slit-lamp microscopy to assess the anterior segment. Assessment of ocular surface status was performed by measuring tear film break-up time (TBUT), corneal fluorescein staining (FSS), and grading conjunctivo

SUMMARY:
Subconjunctival hemorrhage (SCH) is characterized by the rupture of a small conjunctival or episcleral blood vessel, leading to localized extravasation of blood beneath the conjunctiva.1, 2 Non-traumatic cases occur without external mechanical injury.1, 2 Clinically, it manifests as a sharply demarcated bright or dark red patch on the sclera, often prompting concern due to its striking appearance.1 Despite its alarming presentation, SCH is generally a benign condition that neither causes pain nor affects visual acuity, although some patients may report mild ocular discomfort or a foreign-body sensation.1 SCH typically resolves spontaneously within 1 to 2 weeks, analogous to the resolution of a cutaneous bruise, as the extravasated blood is gradually resorbed.3 While most cases are isolated and self-limiting, recurrent SCH or episodes accompanied by other ocular or systemic symptoms warrant further evaluation to exclude underlying systemic disorders.4, 5 Identifying risk factors for SCH is clinically important, as it may facilitate the early diagnosis and management of systemic conditions, thereby reducing the likelihood of recurrence. The most common precipitating factor is minor ocular trauma, such as vigorous eye rubbing.6 Other recognized triggers include acute increases in venous pressure associated with coughing, sneezing, or Valsalva maneuvers, as well as the use of anticoagulant or antiplatelet agents, including warfarin and aspirin.1, 6 Although vascular disorders such as hypertension and diabetes mellitus have been suggested as potential systemic risk factors, the literature addressing these associations remains limited.1, 7, 8 Thus, this study aimed to identify potential risk factors associated with SCH. Initially, a retrospective analysis was conducted to explore candidate risk factors, followed by a prospective study to validate the findings.

DETAILED DESCRIPTION:
a prospective study was performed at Hallym University Kangnam Sacred Heart Hospital, Hallym University Dongtan Sacred Heart Hospital and Hallym University Sacred Heart Hospital from Dec. 2022 to Dec. 2024. Patient assessments included the same systemic variables: sex, diabetes mellitus, hypertension, anticoagulant use (including both antiplatelet agents and novel oral anticoagulants [NOACs]), circulatory agents, and omega-3 supplementation. Circulatory agents included Ginkgo biloba extract formulations such as Gingkomin Tab and Ginexin-F, as well as magnesium, calcium supplements, and vasodilators such as trimetazidine and limaprost.12, 13 Patients were also asked to complete structured questionnaires addressing eye rubbing, sleep deprivation, fatigue, and increased intra-abdominal pressure due to physical factors such as heavy lifting, constipation, coughing, and prone positioning. Ophthalmologic examinations were performed using fundus photography to detect retinal hemorrhages and slit-lamp microscopy to assess the anterior segment. Assessment of ocular surface status was performed by measuring tear film break-up time (TBUT), corneal fluorescein staining (FSS), and grading conjunctivochalasis (CCH).14 TBUT was quantified in seconds based on the interval between the last blink and the first appearance of a dry spot, while FSS was graded using the Oxford grading scale.14 CCH was classified using a modified grading scale based on the number and extent of conjunctival folds. Grade 0 denoted the absence of folds; Grade 1 indicated a single fold; Grade 2 represented multiple folds that did not reach the tear meniscus; and Grade 3 included prominent folds encroaching upon and disrupting the tear meniscus.15

ELIGIBILITY:
Inclusion Criteria:

* The patients aged 19 years or older who visited the ophthalmology outpatient clinic due to non-traumatic subconjunctival hemorrhage and the normal patients who visited the ophthalmology outpatient clinic for an ophthalmological examination were enrolled.

Exclusion Criteria:

* Trauma patients are excluded.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A prospective study was performed at Hallym University Kangnam Sacred Heart Hospital, Hallym University Dongtan Sacred Heart Hospital and Hallym University Sacred Heart Hospital from Dec. 2022 to Dec. 2024. The patients aged 19 years or older who visited the ophthalmology outpatient clinic due to non-traumatic subconjunctival hemorrhage and the normal patients who visited the ophthalmology outpatient clinic for an ophthalmological examination were enrolled. Trauma patients are excluded.
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2022-12-22 (Actual); Primary Completion 2024-12-28 (Actual); Study Completion 2024-12-28 (Actual)

PRIMARY OUTCOMES:
Subconjunctival hemorrhage | From December 2022 to December 2024
  Detection and extent of Subconjunctival hemorrhage

CONTACTS AND LOCATIONS:
Locations (1):
- Hallym University, Kangnam Sacred Heart Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No